CLINICAL TRIAL: NCT03050151
Title: An Open-label, Randomized, Actual Use Study of Dupilumab Auto-injector Device in Patients With Atopic Dermatitis
Brief Title: Study of Dupilumab Auto-injector Device When Used by Patients With Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R668-AD-1607
Record Dates: First submitted 2017-02-08; First posted 2017-02-10 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-05

CONDITIONS: Atopic Disorders; Eczema, Atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (4):
- 1 - Dupilumab (Part A) (Experimental): Dose (dose 1) as per protocol delivered by auto-injector device
  Interventions: Drug: Dupilumab; Device: Auto-injector Device
- 2 - Dupilumab (Part A) (Experimental): Dose (dose 1) as per protocol delivered by prefilled syringe
  Interventions: Drug: Dupilumab; Device: Prefilled syringe
- 3 - Dupilumab (Part B) (Experimental): Dose (dose 2) as per protocol delivered by auto-injector device
  Interventions: Drug: Dupilumab; Device: Auto-injector Device
- 4 - Dupilumab (Part B) (Experimental): Dose (dose 2) as per protocol delivered by prefilled syringe
  Interventions: Drug: Dupilumab; Device: Prefilled syringe

INTERVENTIONS:
Drug: Dupilumab — Administration of dose of Dupilumab as per protocol by auto-injector or prefilled syringe
Device: Auto-injector Device — Delivery of Dupilumab by auto-injector device
  Arms: 1 - Dupilumab (Part A); 3 - Dupilumab (Part B)
Device: Prefilled syringe — Delivery of Dupilumab by prefilled syringe
  Arms: 2 - Dupilumab (Part A); 4 - Dupilumab (Part B)

SUMMARY:
To collect data on actual-use to assess technical performance and user injections of dupilumab auto-injection device by patients with atopic dermatitis (AD).

DETAILED DESCRIPTION:
Study is conducted in 2 parts: part A and part B.

Part A - Patients with moderate-to-severe AD will be randomized to receive dupilumab (dose 1) by auto-injector (AI) device or prefilled syringe.

Once part A is completely enrolled, part B will randomize patients with moderate-to-severe AD to receive dupilumab (dose 2) by auto-injector (AI) device or prefilled syringe.

ELIGIBILITY:
Key Inclusion Criteria:

1. Diagnosis of chronic atopic dermatitis for at least 3 years with inadequate response to topical medications within 6 months before screening
2. Willing and able to comply with all clinic visits and study-related procedures
3. Provide signed informed consent

Key Exclusion Criteria:

1. Patient < 30.0 kilograms (Kg) in weight
2. Patient who has previously participated in a dupilumab clinical study
3. Patient who has been treated with the following:

   * An investigational drug within 8 weeks or within 5 half-lives (if known),whichever is longer, before the baseline visit
   * Immunosuppressive/ immunomodulating drugs (e.g., systemic corticosteroids, cyclosporine, mycophenolate-mufti, IFN-γ, Janus kinase inhibitors, azathioprine, methotrexate, etc.) or Phototherapy for AD within 4 weeks before the baseline visit
   * An experimental monoclonal antibody within 5 half-lives or within 6◦months prior to visit 1 if the half-life is unknown
   * Biologic agents within 5 half-lives (if known) or 16 weeks prior to baseline visit, whichever is longer
   * Anti-immunoglobulin E therapy (omalizumab) within 130 days prior to visit 1
   * A live (attenuated) vaccine within 4 weeks before the baseline visit
4. Patient who has initiated treatment with prescription moisturizers or moisturizers containing additives such as ceramide, hyaluronic acid, urea, or filaggrin degradation products during the screening period (patients may continue using stable doses of such moisturizers if initiated before the screening visit)
5. Patient who has skin comorbidities that may interfere with study assessments
6. Patient with a planned or anticipated major surgical procedure during the patient's participation in this study
7. Women of childbearing potential unwilling to use adequate birth control measures during the study
8. Pregnant or breastfeeding women, or women planning to become pregnant or breastfeed during the study

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2017-11-14 (Actual); Study Completion 2018-02-12 (Actual)

PRIMARY OUTCOMES:
Number of validated AI device-associated product technical failures (PTFs) during the treatment period divided by total number of actual injections | To week 12
Type of validated AI device-associated PTFs during the treatment period divided by total number of actual injections. | To week 12

SECONDARY OUTCOMES:
Number of patients with an AI device-associated PTF | To week 12
Percentage of patients with an AI device-associated PTF | To week 12
Number of AI device-associated product technical complaints (PTCs) divided by total number of actual injections | To week 12
Type of AI device-associated PTCs divided by total number of actual injections | To week 12
Number of patients with an AI device-associated PTC | To week 12
Percentage of patients with an AI device-associated PTC | To week 12
Number of AI device-associated failed drug deliveries (defined as patient failure to administer the full dose at a given attempt, excluding PTF) divided by total number of actual injections | To week 12
Type of AI device-associated failed drug deliveries (defined as patient failure to administer the full dose at a given attempt, excluding PTF) divided by total number of actual injections | To week 12
Number of patients with an AI device-associated failure to deliver dose | To week 12
Percentage of patients with an AI device-associated failure to deliver dose | To week 12
Number of patients with response to patient satisfaction questions with the AI device | To week 12
Percentage of patients with response to patient satisfaction questions with the AI device | To week 12

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (35):
- United States (35):
  - Regeneron Investigational Site, Birmingham, Alabama
  - Regeneron Investigational Site, Fort Smith, Arkansas
  - Regeneron Investigational Site, Long Beach, California
  - Regeneron Investigational Site, Los Angeles, California
  - Regeneron Investigational Site, Murrieta, California
  - Regeneron Investigational Site, Oceanside, California
  - Regeneron Investigational Site, Orange, California
  - Regeneron Investigational Site, Rolling Hills Estates, California
  - Regeneron Investigational Site, Santa Monica, California
  - Regeneron Investigational Site, Denver, Colorado
  - Regeneron Investigational Site, Coral Gables, Florida
  - Regeneron Investigational Site, Tampa, Florida
  - Regeneron Investigational Site, Normal, Illinois
  - Regeneron Investigational Site, Skokie, Illinois
  - Regeneron Investigational Site, Indianapolis, Indiana
  - Regeneron Investigational Site, Rockville, Maryland
  - Regeneron Investigational Site, Plymouth, Minnesota
  - Regeneron Investigational Site, Saint Joseph, Missouri
  - Regeneron Investigational Site, Berlin, New Jersey
  - Regeneron Investigational Site, Windsor, New Jersey
  - Regeneron Investigational Site, Corning, New York
  - Regeneron Investigational Site, Forest Hills, New York
  - Regeneron Investigational Site, New York, New York
  - Regeneron Investigational Site, High Point, North Carolina
  - Regeneron Investigational Site, Raleigh, North Carolina
  - Regeneron Investigational Site, Tulsa, Oklahoma
  - Regeneron Investigational Site, Portland, Oregon
  - Regeneron Investigational Site, Charleston, South Carolina
  - Regeneron Investigational Site, Greer, South Carolina
  - Regeneron Investigational Site, Bellaire, Texas
  - Regeneron Investigational Site, Fort Worth, Texas
  - Regeneron Investigational Site, San Antonio, Texas
  - Regeneron Investigational Site, Webster, Texas
  - Regeneron Investigational Site, Norfolk, Virginia
  - Regeneron Investigational Site, Tacoma, Washington

REFERENCES:
- [Derived] Blauvelt A, Guttman-Yassky E, Paller AS, Simpson EL, Cork MJ, Weisman J, Browning J, Soong W, Sun X, Chen Z, Kosloski MP, Kamal MA, Delevry D, Chuang CC, O'Malley JT, Bansal A. Long-Term Efficacy and Safety of Dupilumab in Adolescents with Moderate-to-Severe Atopic Dermatitis: Results Through Week 52 from a Phase III Open-Label Extension Trial (LIBERTY AD PED-OLE). Am J Clin Dermatol. 2022 May;23(3):365-383. doi: 10.1007/s40257-022-00683-2. Epub 2022 May 14. PMID 35567671